CLINICAL TRIAL: NCT02069938
Title: Brain Computer Interface Control of a Robotic Device
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1312M46742
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Subjects

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Subjects: Noninvasive Brain Computer Interface Control

SUMMARY:
Noninvasive Brain-Computer Interfaces (BCIs) have been used to control a number of virtual and physical objects through the voluntary modulation of brain rhythms. Current issues with noninvasive BCIs include exhausting motor imagery tasks and long training times required to achieve competent control. The investigators will address these issues within this protocol, examining new approaches to reduce the effort required by subjects to control a physical object in the task.

The PI's hypothesis is: Control of a physical robotic device will increase the performance of subjects in BCI tasks that are analogous to virtual tasks due to greater engagement with a physical output.

DETAILED DESCRIPTION:
Subjects will be recruited to participate in controlling a physical robotic device such as a quadcopter or a robotic arm using imagination of movement or other activities as detected by brain waves that can be used to control a robotic device.

The subjects will be able to observe the controlling of a robotics device using one's thought and participate in multiple sessions to learn the skills to better control such a device.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for this study will be healthy, English speaking adult volunteers (18-64 years old).

Exclusion Criteria:

* History of neurological deficit or traumatic brain injury.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects, primarily from individuals on the University of Minnesota Campus and Minneapolis area
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03-13 (Actual); Study Completion 2016-03-13 (Actual)

PRIMARY OUTCOMES:
Percent of trials correct within each session of Brain Computer Interface experiments. | Session 1 through 10, within an average of 5 weeks. Each session separated by at least 24 hours.
  Accuracy and performance metrics of Brain-Computer Interface tasks over time. This will include the percent of trials correct, percent of trials completed, and time to completion within each session. Combining these metrics, we will examine subject learning over sessions with regression. Exact time frame of sessions will be determined by subject and equipment availability.

CONTACTS AND LOCATIONS:
Overall Officials: Bin He, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Nils Hasselmo Hall at the University of Minnesota - Twin Cities Campus, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided